CLINICAL TRIAL: NCT00771615
Title: A Trial to Evaluate the Safety & Immunogenicity of Investigational Influenza Vaccine GSK1557484A in Adults 18-64 Yrs of Age
Brief Title: Immunogenicity & Safety of GSK's Avian Flu Vaccine 1557484A Given to Adults Aged 18-64 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 111729
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: human; Avian; safety; vaccines; influenza; pandemic; immunogenicity; H5N1
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (9):
- A/turkey H5N1 influenza Formulation A Group (Experimental): Subjects previously primed in NCT00510874 study with formulation 1 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation A of GSK A/turkey H5N1 Influenza vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK A/turkey H5N1 Influenza vaccine
- A/turkey H5N1 influenza Formulation B1 Group (Experimental): Subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation B1 of GSK A/turkey H5N1 Influenza vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK A/turkey H5N1 Influenza vaccine
- A/turkey H5N1 influenza Formulation B2 Group (Experimental): Subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation B2 of GSK A/turkey H5N1 Influenza vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK A/turkey H5N1 Influenza vaccine
- A/turkey H5N1 influenza Formulation C1 Group (Experimental): Subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation C1 of GSK A/turkey H5N1 Influenza vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK A/turkey H5N1 Influenza vaccine
- A/turkey H5N1 influenza Formulation C2 Group (Experimental): Subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation C2 of GSK A/turkey H5N1 Influenza vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK A/turkey H5N1 Influenza vaccine
- A/turkey H5N1 influenza Formulation D1 Group (Experimental): Subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation D1 of GSK A/turkey H5N1 Influenza vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK A/turkey H5N1 Influenza vaccine
- A/turkey H5N1 influenza Formulation D2 Group (Experimental): Subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation D2 of GSK A/turkey H5N1 Influenza vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK A/turkey H5N1 Influenza vaccine
- A/turkey H5N1 influenza Formulation E1 Group (Experimental): Subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation E1 of GSK A/turkey H5N1 Influenza vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK A/turkey H5N1 Influenza vaccine
- A/turkey H5N1 influenza Formulation E2 Group (Experimental): Subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation E2 of GSK A/turkey H5N1 Influenza vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK A/turkey H5N1 Influenza vaccine

INTERVENTIONS:
Biological: GSK A/turkey H5N1 Influenza vaccine — One dose administered intramuscularly (IM) in the deltoid region. Different formulations are tested.

SUMMARY:
The purpose of this observer-blind study is to determine whether GSK's avian flu vaccine GSK 1557484A is immunogenic when given to adults aged 18-64 years.

DETAILED DESCRIPTION:
All enrolled subjects will receive 1 dose of study vaccine. All subjects will attend formal study center visits for safety and immunogenicity assessments on Days 0, 10, 42, 84, and 182 with a telephone safety contact on Day 364.

This Protocol Posting has been updated according to Protocol amendment, 8 Dec 08

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults 18 to 64 years of age at time of first vaccination, inclusive.
* Written informed consent obtained from the subject.
* Stable health status as defined by absence of a health event satisfying the definition of a SAE, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within 1 month prior to enrollment.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line, or mobile, but NOT a pay phone or other multiple-user device.
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.
* Subjects who the investigator believes can and will comply with the requirements of the protocol.

Exclusion Criteria:

* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if clinically stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Presence of an oral temperature >= 37.8ºC, or acute symptoms greater than "mild" severity on the scheduled date of vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition including history of human immunodeficiency virus (HIV) infection.
* Receipt of systemic glucocorticoids (prednisone >= 10 mg/day for more than 14 consecutive days) within 1 month prior to study enrollment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 weeks of receipt of seasonal influenza vaccine.
* Any significant disorder of coagulation or treatment with Coumadin derivatives or heparin.
* Administration of any vaccines within 30 days before the first study vaccine dose.
* Previous administration of any H5N1 vaccine.
* Use of any investigational or non-registered product (drug or vaccine) or planned participation in another investigational study within 30 days prior to study enrollment, or during the 12 months following test article administration. Use of any investigational or non-registered product with immunosuppressive properties is exclusionary at any time during the trial.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrollment or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-hCG) test result prior to vaccination.
* Lactating or nursing.
* Women of child bearing potential (who lack a history of reliable contraceptive practices. The provision of this history does NOT replace the requirement to perform, and obtain negative results in pregnancy urine tests prior to vaccination.
* Known receipt of analgesic or antipyretic medication with the specific intent of prophylaxis of vaccine reactogenicity on the day of vaccination. Subjects on stable chronic regimens of potentially analgesic or anti-pyretic medications for pre-existing diagnoses are not required to discontinue them.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 469 (Actual)
Dates: Start 2008-10-16; Primary Completion 2009-05-26 (Actual); Study Completion 2009-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (7):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Las Vegas, Nevada
- Canada (3):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Risi G, Frenette L, Langley JM, Li P, Riff D, Sheldon E, Vaughn DW, Fries L. Immunological priming induced by a two-dose series of H5N1 influenza antigen, administered alone or in combination with two different formulations of AS03 adjuvant in adults: results of a randomised single heterologous booster dose study at 15 months. Vaccine. 2011 Aug 26;29(37):6408-18. doi: 10.1016/j.vaccine.2011.04.072. Epub 2011 May 7. PMID 21554915
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111729 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111729 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111729 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111729 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111729 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111729 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111729 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A/Turkey H5N1 Influenza Formulation A Group | A/Turkey H5N1 Influenza Formulation B1 Group | A/Turkey H5N1 Influenza Formulation B2 Group | A/Turkey H5N1 Influenza Formulation C1 Group | A/Turkey H5N1 Influenza Formulation C2 Group | A/Turkey H5N1 Influenza Formulation D1 Group | A/Turkey H5N1 Influenza Formulation D2 Group | A/Turkey H5N1 Influenza Formulation E1 Group | A/Turkey H5N1 Influenza Formulation E2 Group
Started | 49 | 72 | 41 | 60 | 40 | 61 | 46 | 59 | 41
Completed | 48 (Up to Day 364) | 70 (Up to Day 364) | 40 (Up to Day 364) | 59 (Up to Day 364) | 40 (Up to Day 364) | 60 (Up to Day 364) | 45 (Up to Day 364) | 58 (Up to Day 364) | 41 (Up to Day 364)
Not Completed | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A/Turkey H5N1 Influenza Formulation A Group | A/Turkey H5N1 Influenza Formulation B1 Group | A/Turkey H5N1 Influenza Formulation B2 Group | A/Turkey H5N1 Influenza Formulation C1 Group | A/Turkey H5N1 Influenza Formulation C2 Group | A/Turkey H5N1 Influenza Formulation D1 Group | A/Turkey H5N1 Influenza Formulation D2 Group | A/Turkey H5N1 Influenza Formulation E1 Group | A/Turkey H5N1 Influenza Formulation E2 Group | Total
Number analyzed (Participants) | 49 | 72 | 41 | 60 | 40 | 61 | 46 | 59 | 41 | 469
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (11.47) | 40.6 (12.02) | 41.1 (11.82) | 41.2 (12.33) | 41.1 (12.46) | 42.4 (11.15) | 41.2 (9.78) | 40.6 (12.01) | 41.6 (11.60) | 41.3 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 42 | 20 | 38 | 21 | 40 | 31 | 37 | 19 | 277
  Male | 20 | 30 | 21 | 22 | 19 | 21 | 15 | 22 | 22 | 192

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination (Day 0) titer less than (<) 1:10 for HI and a post-vaccination reciprocal titer greater than or equal to (≥) 1:40, or a pre-vaccination reciprocal titer ≥ 1:10 for HI and at least a 4-fold increase in post-vaccination reciprocal titer.
Time Frame: At Day 10
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom a complete set of immunogenicity data required for the primary endpoint were available.
Measure: Count of Participants; unit: Participants
Groups:
- A/Turkey H5N1 Influenza A Group: Subjects previously primed in NCT00510874 study with formulation 1 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation A of GSK A/turkey H5N1 Influenza vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- A/Turkey H5N1 Influenza B1 + D1 Group: Subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation B1 of GSK A/turkey H5N1 Influenza vaccine and subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation D1 of GSK A/turkey H5N1 Influenza vaccine; data for both groups are pooled.
  The different formulations of GSK A/turkey H5N1 Influenza vaccine were administered intramuscularly in the deltoid region of the non-dominant arm.
- A/Turkey H5N1 Influenza C1 + E1 Group: Subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation C1 of GSK A/turkey H5N1 Influenza vaccine and subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation E1 of GSK A/turkey H5N1 Influenza vaccine; data for both groups are pooled.
  The different formulations of GSK A/turkey H5N1 Influenza vaccine were administered intramuscularly in the deltoid region of the non-dominant arm.
- A/Turkey H5N1 Influenza B2 + D2 Group: Subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation B2 of GSK A/turkey H5N1 Influenza vaccine and subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation D2 of GSK A/turkey H5N1 Influenza vaccine; data for both groups are pooled.
  The different formulations of GSK A/turkey H5N1 Influenza vaccine were administered intramuscularly in the deltoid region of the non-dominant arm.
- A/Turkey H5N1 Influenza C2 + E2 Group: Subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation C2 of GSK A/turkey H5N1 Influenza vaccine and subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation E2 of GSK A/turkey H5N1 Influenza vaccine; data for both groups are pooled.
  The different formulations of GSK A/turkey H5N1 Influenza vaccine were administered intramuscularly in the deltoid region of the non-dominant arm.
- A/Turkey H5N1 Influenza B1 + C1 Group: Subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation B1 of GSK A/turkey H5N1 Influenza vaccine and subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation C1 of GSK A/turkey H5N1 Influenza vaccine; data for both groups are pooled.
  The different formulations of GSK A/turkey H5N1 Influenza vaccine were administered intramuscularly in the deltoid region of the non-dominant arm.
- A/Turkey H5N1 Influenza D1 + E1 Group: Subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation D1 of GSK A/turkey H5N1 Influenza vaccine and subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation E1 of GSK A/turkey H5N1 Influenza vaccine; data for both groups are pooled.
  The different formulations of GSK A/turkey H5N1 Influenza vaccine were administered intramuscularly in the deltoid region of the non-dominant arm.
- A/Turkey H5N1 Influenza B2 + C2 Group: Subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation B2 of GSK A/turkey H5N1 Influenza vaccine and subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (Q-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation C2 of GSK A/turkey H5N1 Influenza vaccine; data for both groups are pooled.
  The different formulations of GSK A/turkey H5N1 Influenza vaccine were administered intramuscularly in the deltoid region of the non-dominant arm.
- A/Turkey H5N1 Influenza D2 + E2 Group: Subjects previously primed in NCT00510874 study with formulation 2 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation D2 of GSK A/turkey H5N1 Influenza vaccine and subjects previously primed in NCT00510874 study with formulation 3 of Influenza A (D-Pan H5N1) virus monovalent vaccine (A/Indonesia) were boosted with a single dose of formulation E2 of GSK A/turkey H5N1 Influenza vaccine; data for both groups are pooled.
  The different formulations of GSK A/turkey H5N1 Influenza vaccine were administered intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
Participants | 43 | 121 | 109 | 57 | 56 | 122 | 108 | 51 | 62

2. Primary Outcome: Number of Subjects Seroprotected for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain
Description: A seroprotected subject against the A/turkey virus strain was defined as a subject with serum HI antibody reciprocal titer ≥ 1:40 post-vaccination, a level of HI antibodies that may correlate with benefit in protection against influenza.
Time Frame: At Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
Participants | 44 | 125 | 113 | 76 | 67 | 127 | 111 | 69 | 74

3. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: HI antibody titers were expressed as geometric mean titers (GMTs). The cut-off of the assay was the seropositivity cut-off of ≥ 1:10.
Time Frame: At Day 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
Titer | 229.6 [148.6 to 354.9] | 847.3 [686.1 to 1046.4] | 810.5 [666.6 to 985.3] | 121.9 [89.7 to 165.7] | 86.9 [64.7 to 116.7] | 838.5 [703.1 to 1000.1] | 819.8 [647.8 to 1037.3] | 97.9 [70.3 to 136.4] | 108.6 [82.3 to 143.3]

4. Secondary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strains.
Description: as for outcome 1
Time Frame: At Day 0 to Day 42 and at Day 0 to Day 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 128 | 113 | 85 | 80 | 129 | 112 | 79 | 86
Participants
  A/turkey, D 42 | 41 | 123 | 108 | 55 | 51 | 123 | 108 | 45 | 61
  A/turkey, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/turkey, D 182 | 28 | 105 | 90 | 38 | 38 | 103 | 92 | 31 | 45

5. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the A/Turkey/Turkey/1/2005 Virus Strain.
Description: Titers were expressed as geometric mean titers (GMTs). The cut-off of the assay was the seropositivity cut-off of ≥ 1:10
Time Frame: At Day 0, Day 10, Day 42 and Day 182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 128 | 113 | 85 | 80 | 129 | 112 | 79 | 86
Titer
  A/turkey, D 0 | 6.1 [5.0 to 7.5] | 13.5 [11.3 to 16.3] | 14.4 [11.6 to 18.0] | 14.2 [11.3 to 17.9] | 10.9 [8.7 to 13.6] | 14.1 [11.6 to 17.2] | 13.7 [11.1 to 16.9] | 13.2 [10.3 to 17.1] | 11.8 [9.6 to 14.5]
  A/turkey, D 10: number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/turkey, D 10 | 229.6 [148.6 to 354.9] | 847.3 [686.1 to 1046.4] | 810.5 [666.6 to 985.3] | 121.9 [89.7 to 165.7] | 86.9 [64.7 to 116.7] | 838.5 [703.1 to 1000.1] | 819.8 [647.8 to 1037.3] | 97.9 [70.3 to 136.4] | 108.6 [82.3 to 143.3]
  A/turkey, D 42 | 155.4 [102.1 to 236.3] | 652.2 [525.3 to 809.8] | 699.5 [561.9 to 870.8] | 126.3 [91.6 to 174.1] | 81.4 [59.6 to 111.2] | 653.9 [545.5 to 783.9] | 697.8 [539.2 to 903.2] | 90.9 [64.7 to 127.6] | 113.6 [84.1 to 153.4]
  A/turkey, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/turkey, D 182 | 40.9 [26.8 to 62.4] | 221.5 [172.3 to 284.6] | 238.4 [185.1 to 307.0] | 62.7 [44.9 to 87.5] | 42.9 [31.6 to 58.3] | 213.3 [170.5 to 266.9] | 249.1 [187.6 to 330.8] | 51.1 [37.2 to 70.3] | 53.2 [38.3 to 73.8]

6. Secondary Outcome: HI Antibody Geometric Mean Fold Rise (GMFR) Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: GMFR were defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the Day 0 reciprocal HI titer.
Time Frame: At Day 0 to Day 10, Day 42 and Day 182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 128 | 113 | 85 | 80 | 129 | 112 | 79 | 86
fold change
  A/turkey, D 10: number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/turkey, D 10 | 37.4 [23.3 to 59.9] | 61.6 [47.4 to 80.1] | 56.3 [43.5 to 72.8] | 8.5 [6.0 to 12.1] | 8.0 [6.0 to 10.7] | 58.4 [45.5 to 74.9] | 59.8 [45.5 to 78.6] | 7.4 [5.2 to 10.5] | 9.1 [6.8 to 12.3]
  A/turkey, D 42 | 25.3 [16.6 to 38.5] | 48.2 [37.2 to 62.5] | 48.6 [37.5 to 63.0] | 8.9 [6.2 to 12.9] | 7.5 [5.6 to 10.1] | 46.3 [36.2 to 59.2] | 50.9 [38.6 to 67.1] | 6.9 [4.8 to 9.8] | 9.6 [7.1 to 13.1]
  A/turkey, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/turkey, D 182 | 6.7 [4.4 to 10.0] | 16.4 [12.4 to 21.5] | 16.6 [12.7 to 21.6] | 4.4 [3.0 to 6.3] | 3.9 [2.9 to 5.2] | 15.1 [11.6 to 19.6] | 18.2 [13.7 to 24.1] | 3.9 [2.7 to 5.4] | 4.4 [3.2 to 6.1]

7. Secondary Outcome: HI Antibody Titers Against the A/Indonesia/5/2005 (A/Indo) Virus Strain.
Description: as for outcome 5
Time Frame: At Day 0, Day 10, Day 42 and Day 182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 128 | 113 | 85 | 80 | 129 | 112 | 79 | 86
Titer
  A/Indo, D 0 | 7.3 [5.6 to 9.4] | 26.1 [20.8 to 32.7] | 23.8 [18.6 to 30.5] | 25.5 [19.3 to 33.7] | 18.5 [13.9 to 24.5] | 25.5 [20.2 to 32.1] | 24.5 [19.2 to 31.1] | 22.0 [16.6 to 29.1] | 21.7 [16.3 to 28.8]
  A/Indo, D 10: number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/Indo, D 10 | 286.5 [187.6 to 437.5] | 905.0 [743.7 to 1101.4] | 888.6 [739.6 to 1067.5] | 176.7 [131.9 to 236.8] | 113.6 [83.2 to 155.1] | 873.5 [738.5 to 1033.3] | 924.9 [745.0 to 1148.1] | 124.6 [89.4 to 173.8] | 161.3 [122.3 to 212.8]
  A/Indo, D 42 | 192.3 [129.3 to 286.1] | 740.8 [604.7 to 907.4] | 798.1 [656.6 to 970.1] | 168.7 [123.5 to 230.5] | 108.8 [77.7 to 152.4] | 728.1 [613.5 to 864.1] | 814.6 [646.3 to 1026.8] | 107.8 [75.6 to 153.8] | 169.3 [126.1 to 227.2]
  A/Indo, D182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/Indo, D182 | 34.8 [22.6 to 53.6] | 213.8 [166.4 to 274.6] | 224.2 [174.4 to 288.3] | 58.7 [41.2 to 83.6] | 38.6 [28.0 to 53.3] | 197.3 [156.0 to 249.5] | 246.0 [188.0 to 321.9] | 42.7 [30.4 to 60.0] | 53.4 [37.9 to 75.2]

8. Secondary Outcome: Number of Subjects Seroprotected for Haemagglutination Inhibition (HI) Antibodies Against the A/Indonesia/5/2005 (A/Indo) and A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strains.
Description: A seroprotected subject was defined as a subject with serum HI antibody reciprocal titer ≥ 1:40 post-vaccination, a level of HI antibodies that may correlate with benefit in protection against influenza.
Time Frame: At Day 0, Day 10, Day 42 and Day 182 for A/Indo and at Day 0, Day 42 and Day 182 for A/turkey virus strains.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 128 | 113 | 85 | 80 | 129 | 112 | 79 | 86
Participants
  A/Indo, D 0 | 5 | 70 | 56 | 44 | 31 | 68 | 58 | 34 | 41
  A/Indo, D 10: number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/Indo, D 10 | 44 | 125 | 113 | 79 | 68 | 127 | 111 | 69 | 78
  A/Indo, D 42 | 44 | 126 | 113 | 78 | 67 | 129 | 110 | 66 | 79
  A/Indo, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/Indo, D 182 | 28 | 116 | 106 | 58 | 47 | 121 | 101 | 48 | 57
  A/turkey, D 0 | 3 | 32 | 35 | 25 | 16 | 36 | 31 | 23 | 18
  A/turkey, D 42 | 41 | 126 | 113 | 74 | 62 | 129 | 110 | 64 | 72
  A/turkey, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/turkey, D 182 | 31 | 119 | 106 | 58 | 53 | 122 | 103 | 54 | 57

9. Secondary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Indonesia/5/2005 (A/Indo) Virus Strains.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer less than (<) 1:10 and a post-vaccination reciprocal titer greater than or equal to (≥) 1:40 or a pre-vaccination reciprocal titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Day 0 to Day 10, Day 42 and Day 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 128 | 113 | 85 | 80 | 129 | 112 | 79 | 86
Participants
  A/Indo, D 10: number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/Indo, D 10 | 42 | 122 | 108 | 50 | 44 | 122 | 108 | 41 | 53
  A/Indo, D 42 | 42 | 120 | 105 | 48 | 43 | 121 | 104 | 38 | 53
  A/Indo, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/Indo, D 182 | 25 | 91 | 84 | 24 | 22 | 96 | 79 | 20 | 26

10. Secondary Outcome: HI Antibody Geometric Mean Fold Rise (GMFR) Against the A/Indonesia/5/2005 (A/Indo) Virus Strains.
Description: as for outcome 6
Time Frame: At Day 10, Day 42 and Day 182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 128 | 113 | 85 | 80 | 129 | 112 | 79 | 86
fold change
  A/Indo, D 10: number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/Indo, D 10 | 39.3 [24.8 to 62.4] | 34.7 [26.8 to 44.8] | 37.3 [28.5 to 48.8] | 6.8 [4.9 to 9.5] | 6.1 [4.5 to 8.3] | 34.3 [26.8 to 43.8] | 37.8 [28.5 to 50.2] | 5.7 [4.1 to 7.9] | 7.3 [5.4 to 10.0]
  A/Indo, D 42 | 26.4 [17.2 to 40.5] | 28.4 [22.0 to 36.7] | 33.5 [25.4 to 44.3] | 6.6 [4.7 to 9.4] | 5.9 [4.3 to 8.1] | 28.6 [22.3 to 36.6] | 33.3 [24.9 to 44.5] | 4.9 [3.4 to 7.0] | 7.8 [5.7 to 10.7]
  A/Indo, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/Indo, D 182 | 4.8 [3.1 to 7.4] | 8.2 [6.3 to 10.7] | 9.4 [7.2 to 12.3] | 2.3 [1.6 to 3.3] | 2.1 [1.6 to 2.8] | 7.7 [6.0 to 9.9] | 10.1 [7.6 to 13.4] | 1.9 [1.4 to 2.7] | 2.5 [1.8 to 3.4]

11. Secondary Outcome: Microneutralization (MN) Antibody Titers Against the A/Turkey/Turkey/1/2005 (A/Turkey), A/Indonesia/5/2005 (A/Indo) and A/Vietnam/1194/2004 (A/Vie) Virus Strains.
Description: MN antibody titers were expressed as geometric mean titers (GMTs). The cut-off of the assay was the seropositivity cut-off of ≥ 1:28.
Time Frame: At Day 0, Day 10, Day 42 and Day 182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 128 | 113 | 85 | 80 | 129 | 112 | 79 | 86
Titer
  A/turkey, D 0 | 27.5 [20.6 to 36.7] | 115.4 [92.7 to 143.7] | 114.6 [91.0 to 144.4] | 102.9 [82.4 to 128.4] | 94.9 [71.0 to 126.9] | 115.0 [92.4 to 143.2] | 115.1 [91.3 to 145.0] | 95.9 [73.8 to 124.6] | 101.9 [79.2 to 130.9]
  A/turkey, D 10: number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/turkey, D 10 | 2211.5 [1579.1 to 3097.1] | 5367.7 [4604.3 to 6257.6] | 5191.4 [4403.4 to 6120.5] | 1276.2 [962.5 to 1692.1] | 976.0 [740.6 to 1286.1] | 5670.5 [4958.4 to 6484.8] | 4876.8 [4057.3 to 5861.7] | 1026.9 [756.6 to 1393.9] | 1213.4 [939.3 to 1567.5]
  A/turkey, D 42: number analyzed (Participants) | 47 | 128 | 113 | 85 | 79 | 129 | 112 | 79 | 85
  A/turkey, D 42 | 1582.9 [1080.4 to 2319.0] | 4777.7 [4037.3 to 5654.0] | 4649.4 [3884.9 to 5564.3] | 1261.2 [950.0 to 1674.2] | 906.0 [673.6 to 1218.6] | 4915.6 [4212.6 to 5735.8] | 4498.4 [3699.9 to 5469.2] | 935.7 [688.9 to 1271.0] | 1223.9 [929.0 to 1612.3]
  A/turkey, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/turkey, D 182 | 349.7 [246.2 to 496.7] | 1509.9 [1230.5 to 1852.8] | 1484.8 [1181.6 to 1865.8] | 471.5 [352.2 to 631.3] | 342.2 [254.8 to 459.7] | 1375.0 [1123.6 to 1682.7] | 1653.6 [1313.4 to 2081.9] | 332.3 [245.2 to 450.3] | 484.8 [365.7 to 642.8]
  A/Indo, D 0 | 72.8 [52.0 to 101.9] | 326.0 [280.2 to 379.3] | 300.2 [256.7 to 351.1] | 343.4 [288.8 to 408.2] | 262.0 [220.9 to 310.9] | 308.1 [263.0 to 361.0] | 320.1 [276.3 to 371.0] | 288.1 [238.3 to 348.3] | 313.7 [267.3 to 368.2]
  A/Indo, D 10: number analyzed (Participants) | 47 | 126 | 113 | 85 | 80 | 127 | 112 | 79 | 85
  A/Indo, D 10 | 2311.5 [1708.9 to 3126.5] | 5807.1 [5144.8 to 6554.7] | 5680.0 [4943.7 to 6525.9] | 1516.5 [1194.5 to 1925.3] | 1250.0 [1002.6 to 1558.5] | 6011.0 [5424.1 to 6661.5] | 5460.9 [4670.2 to 6385.4] | 1240.9 [966.2 to 1593.7] | 1523.4 [1233.4 to 1881.5]
  A/Indo, D 42 | 1622.0 [1105.2 to 2380.4] | 5080.1 [4412.0 to 5849.3] | 5054.1 [4276.6 to 5972.8] | 1537.2 [1192.0 to 1982.3] | 1194.5 [940.0 to 1517.9] | 5157.1 [4518.4 to 5886.0] | 4967.0 [4163.2 to 5926.0] | 1178.0 [916.6 to 1514.0] | 1552.4 [1216.5 to 1981.0]
  A/Indo, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/Indo, D 182 | 380.8 [267.5 to 542.1] | 1482.3 [1223.3 to 1796.1] | 1556.0 [1265.4 to 1913.3] | 535.5 [416.8 to 688.0] | 378.4 [288.7 to 496.1] | 1358.2 [1130.0 to 1632.5] | 1721.5 [1390.0 to 2132.1] | 379.4 [287.9 to 500.0] | 534.2 [417.9 to 682.8]
  A/Vie, D 0 | 181.3 [138.5 to 237.4] | 210.1 [177.0 to 249.4] | 249.0 [217.8 to 284.7] | 197.3 [159.0 to 244.9] | 205.5 [161.8 to 261.1] | 237.5 [206.4 to 273.2] | 216.5 [181.6 to 258.2] | 198.7 [155.2 to 254.3] | 203.7 [165.2 to 251.0]
  A/Vie, D 10: number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/Vie, D 10 | 662.5 [526.4 to 833.9] | 1564.1 [1312.0 to 1864.7] | 1350.1 [1142.2 to 1595.8] | 552.0 [447.8 to 680.4] | 430.5 [351.8 to 527.0] | 1485.0 [1250.8 to 1763.1] | 1430.0 [1202.3 to 1700.8] | 509.3 [408.1 to 635.6] | 470.8 [387.7 to 571.8]
  A/Vie, D 42 | 529.3 [426.2 to 657.2] | 1213.8 [1004.5 to 1466.6] | 1249.3 [1033.4 to 1510.3] | 589.4 [469.5 to 739.9] | 377.8 [311.3 to 458.5] | 1168.1 [969.8 to 1407.1] | 1306.0 [1076.8 to 1584.1] | 481.8 [382.4 to 607.0] | 469.0 [381.8 to 576.2]
  A/Vie, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/Vie, D 182 | 112.5 [84.5 to 149.8] | 432.5 [366.6 to 510.2] | 324.9 [260.0 to 406.1] | 172.7 [137.9 to 216.3] | 144.1 [119.9 to 173.3] | 371.4 [309.2 to 446.1] | 386.3 [313.8 to 475.5] | 151.7 [120.5 to 191.0] | 164.5 [136.7 to 198.1]

12. Secondary Outcome: Number of Subjects Seropositive for MN Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey), A/Indonesia/5/2005 (A/Indo) and A/Vietnam/1194/2004 (A/Vie) Virus Strains.
Description: A seropositive subject was defined as a vaccinated subject who had a MN antibody titer ≥ the cut-off value of 1:28.
Time Frame: At Day 0, Day 10, Day 42 and Day 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 128 | 113 | 85 | 80 | 129 | 112 | 79 | 86
Participants
  A/turkey, D 0 | 20 | 116 | 102 | 80 | 68 | 114 | 104 | 71 | 77
  A/turkey, D 10: number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/turkey, D 10 | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/turkey, D 42: number analyzed (Participants) | 47 | 128 | 113 | 85 | 79 | 129 | 112 | 79 | 85
  A/turkey, D 42 | 47 | 128 | 113 | 85 | 79 | 129 | 112 | 79 | 85
  A/turkey, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/turkey, D 182 | 46 | 128 | 111 | 82 | 77 | 127 | 112 | 75 | 84
  A/Indo, D 0 | 36 | 126 | 112 | 85 | 79 | 127 | 111 | 78 | 86
  A/Indo, D 10: number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/Indo, D 10 | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/Indo, D 42 | 46 | 128 | 113 | 85 | 80 | 129 | 112 | 79 | 86
  A/Indo, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/Indo, D 182 | 46 | 128 | 112 | 83 | 78 | 128 | 112 | 78 | 83
  A/Vie, D 0 | 46 | 120 | 112 | 80 | 76 | 126 | 106 | 73 | 83
  A/Vie, D10: number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/Vie, D10 | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
  A/Vie, D 42 | 47 | 128 | 112 | 85 | 80 | 128 | 112 | 79 | 86
  A/Vie, D 182: number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
  A/Vie, D 182 | 44 | 126 | 106 | 80 | 77 | 124 | 108 | 74 | 83

13. Secondary Outcome: Vaccine Response Rate (VRR) for Microneutralization (MN) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey), A/Indonesia/5/2005 (A/Indo) and A/Vietnam/1194/2004 (A/Vie) Virus Strains.
Description: VRR was defined as a 4-fold rise from a detectable baseline titer or a rise from undetectable (< 1:28, recorded 1:14 if < 1:28) to ≥ 1:56 in the subjects.
Time Frame: At Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 126 | 113 | 84 | 80 | 127 | 112 | 79 | 85
Participants
  A/turkey, Day 10 | 46 | 122 | 112 | 66 | 56 | 124 | 110 | 55 | 67
  A/Indo, Day 10 | 45 | 121 | 105 | 36 | 40 | 122 | 104 | 32 | 44
  A/Vie, Day 10 | 19 | 84 | 64 | 29 | 18 | 75 | 73 | 24 | 23

14. Secondary Outcome: Vaccine Response Rate (VRR) for Microneutralization (MN) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey), A/Indonesia/5/2005 (A/Indo) and A/Vietnam/1194/2004 (A/Vie) Virus Strains
Description: as for outcome 13
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 128 | 113 | 85 | 80 | 129 | 112 | 79 | 86
Participants
  A/turkey, Day 42: number analyzed (Participants) | 47 | 128 | 113 | 85 | 79 | 129 | 112 | 79 | 85
  A/turkey, Day 42 | 46 | 121 | 110 | 67 | 58 | 122 | 109 | 56 | 69
  A/Indo, D 42 | 41 | 118 | 103 | 39 | 38 | 119 | 102 | 31 | 46
  A/Vie, D 42 | 15 | 73 | 65 | 32 | 15 | 71 | 67 | 25 | 22

15. Secondary Outcome: Vaccine Response Rate (VRR) for Microneutralization (MN) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey), A/Indonesia/5/2005 (A/Indo) and A/Vietnam/1194/2004 (A/Vie) Virus Strains.
Description: as for outcome 13
Time Frame: At Day 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza A Group | A/Turkey H5N1 Influenza B1 + D1 Group | A/Turkey H5N1 Influenza C1 + E1 Group | A/Turkey H5N1 Influenza B2 + D2 Group | A/Turkey H5N1 Influenza C2 + E2 Group | A/Turkey H5N1 Influenza B1 + C1 Group | A/Turkey H5N1 Influenza D1 + E1 Group | A/Turkey H5N1 Influenza B2 + C2 Group | A/Turkey H5N1 Influenza D2 + E2 Group
Number analyzed (Participants) | 47 | 128 | 113 | 84 | 79 | 129 | 112 | 79 | 84
Participants
  A/turkey, Day 182 | 34 | 103 | 89 | 43 | 36 | 102 | 90 | 35 | 44
  A/Indo, Day 182 | 28 | 68 | 72 | 15 | 17 | 71 | 69 | 13 | 19
  A/Vie, Day 182 | 5 | 32 | 22 | 11 | 5 | 24 | 30 | 7 | 9

16. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any solicited local symptoms regardless of their intensity grade.
Time Frame: Within the 7-day (Days 0-6) post vaccination period.
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received study vaccine and for whom any post-vaccination data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza Formulation A Group | A/Turkey H5N1 Influenza Formulation B1 Group | A/Turkey H5N1 Influenza Formulation B2 Group | A/Turkey H5N1 Influenza Formulation C1 Group | A/Turkey H5N1 Influenza Formulation C2 Group | A/Turkey H5N1 Influenza Formulation D1 Group | A/Turkey H5N1 Influenza Formulation D2 Group | A/Turkey H5N1 Influenza Formulation E1 Group | A/Turkey H5N1 Influenza Formulation E2 Group
Number analyzed (Participants) | 49 | 72 | 40 | 60 | 40 | 60 | 46 | 58 | 41
Participants
  Any Pain | 41 | 59 | 9 | 53 | 10 | 48 | 13 | 46 | 6
  Any Redness | 1 | 3 | 0 | 4 | 0 | 4 | 0 | 1 | 0
  Any Swelling | 6 | 2 | 0 | 4 | 0 | 5 | 1 | 2 | 0

17. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited General Symptoms.
Description: Solicited general symptoms assessed were fatigue, headache, joint pain at other location (joint pain), muscle aches, shivering, sweating and fever. Any =occurrence of any solicited general symptoms reported irrespective of intensity grade and relationship to vaccination. Any fever = oral temperature ≥ 38.0 degrees Celsius (°C).
Time Frame: Within the 7-day (Days 0-6) post vaccination period.
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza Formulation A Group | A/Turkey H5N1 Influenza Formulation B1 Group | A/Turkey H5N1 Influenza Formulation B2 Group | A/Turkey H5N1 Influenza Formulation C1 Group | A/Turkey H5N1 Influenza Formulation C2 Group | A/Turkey H5N1 Influenza Formulation D1 Group | A/Turkey H5N1 Influenza Formulation D2 Group | A/Turkey H5N1 Influenza Formulation E1 Group | A/Turkey H5N1 Influenza Formulation E2 Group
Number analyzed (Participants) | 49 | 72 | 40 | 60 | 40 | 60 | 46 | 58 | 41
Participants
  Any Fatigue | 10 | 18 | 3 | 20 | 6 | 18 | 4 | 23 | 11
  Any Headache | 11 | 22 | 4 | 25 | 5 | 17 | 8 | 17 | 10
  Any Joint pain | 5 | 16 | 1 | 10 | 4 | 12 | 2 | 19 | 4
  Any Muscle aches | 10 | 29 | 3 | 17 | 7 | 21 | 8 | 28 | 8
  Any Shivering | 3 | 9 | 1 | 8 | 0 | 7 | 1 | 9 | 2
  Any Sweating | 4 | 4 | 0 | 5 | 0 | 3 | 1 | 6 | 2
  Any Fever | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 4 | 0

18. Secondary Outcome: Number of Subjects With Medically-attended Adverse Events (MAEs).
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Any was defined as any occurrence of MAE(s).
Time Frame: From Day 0 to Day 378
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza Formulation A Group | A/Turkey H5N1 Influenza Formulation B1 Group | A/Turkey H5N1 Influenza Formulation B2 Group | A/Turkey H5N1 Influenza Formulation C1 Group | A/Turkey H5N1 Influenza Formulation C2 Group | A/Turkey H5N1 Influenza Formulation D1 Group | A/Turkey H5N1 Influenza Formulation D2 Group | A/Turkey H5N1 Influenza Formulation E1 Group | A/Turkey H5N1 Influenza Formulation E2 Group
Number analyzed (Participants) | 49 | 72 | 41 | 60 | 40 | 61 | 46 | 59 | 41
Participants | 17 | 24 | 13 | 18 | 13 | 21 | 16 | 20 | 10

19. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms."Any" was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: From Day 0 to Day 42
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza Formulation A Group | A/Turkey H5N1 Influenza Formulation B1 Group | A/Turkey H5N1 Influenza Formulation B2 Group | A/Turkey H5N1 Influenza Formulation C1 Group | A/Turkey H5N1 Influenza Formulation C2 Group | A/Turkey H5N1 Influenza Formulation D1 Group | A/Turkey H5N1 Influenza Formulation D2 Group | A/Turkey H5N1 Influenza Formulation E1 Group | A/Turkey H5N1 Influenza Formulation E2 Group
Number analyzed (Participants) | 49 | 72 | 41 | 60 | 40 | 61 | 46 | 59 | 41
Participants | 9 | 27 | 12 | 26 | 11 | 21 | 12 | 23 | 9

20. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs).
Description: A SAE was defined as any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination.
Time Frame: From Day 0 to Day 378
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | A/Turkey H5N1 Influenza Formulation A Group | A/Turkey H5N1 Influenza Formulation B1 Group | A/Turkey H5N1 Influenza Formulation B2 Group | A/Turkey H5N1 Influenza Formulation C1 Group | A/Turkey H5N1 Influenza Formulation C2 Group | A/Turkey H5N1 Influenza Formulation D1 Group | A/Turkey H5N1 Influenza Formulation D2 Group | A/Turkey H5N1 Influenza Formulation E1 Group | A/Turkey H5N1 Influenza Formulation E2 Group
Number analyzed (Participants) | 49 | 72 | 41 | 60 | 40 | 61 | 46 | 59 | 41
Participants | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs): During the entire study period i.e. Day 0 to Day 378; Systematically assessed adverse events (AEs): During the 7-day (Days 0-6) post vaccination period. Non-systematically assessed AE: During Days 0 - 42.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | A/Turkey H5N1 Influenza Formulation A Group | A/Turkey H5N1 Influenza Formulation B1 Group | A/Turkey H5N1 Influenza Formulation B2 Group | A/Turkey H5N1 Influenza Formulation C1 Group | A/Turkey H5N1 Influenza Formulation C2 Group | A/Turkey H5N1 Influenza Formulation D1 Group | A/Turkey H5N1 Influenza Formulation D2 Group | A/Turkey H5N1 Influenza Formulation E1 Group | A/Turkey H5N1 Influenza Formulation E2 Group
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/72 | 1/41 | 1/60 | 3/40 | 1/61 | 1/46 | 0/59 | 0/41
Other Adverse Events (participants affected / at risk) | 45/49 | 60/72 | 15/41 | 54/60 | 19/40 | 52/61 | 21/46 | 51/59 | 21/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A/Turkey H5N1 Influenza Formulation A Group (N=49) | A/Turkey H5N1 Influenza Formulation B1 Group (N=72) | A/Turkey H5N1 Influenza Formulation B2 Group (N=41) | A/Turkey H5N1 Influenza Formulation C1 Group (N=60) | A/Turkey H5N1 Influenza Formulation C2 Group (N=40) | A/Turkey H5N1 Influenza Formulation D1 Group (N=61) | A/Turkey H5N1 Influenza Formulation D2 Group (N=46) | A/Turkey H5N1 Influenza Formulation E1 Group (N=59) | A/Turkey H5N1 Influenza Formulation E2 Group (N=41)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug abuse (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | A/Turkey H5N1 Influenza Formulation A Group (N=49) | A/Turkey H5N1 Influenza Formulation B1 Group (N=72) | A/Turkey H5N1 Influenza Formulation B2 Group (N=41) | A/Turkey H5N1 Influenza Formulation C1 Group (N=60) | A/Turkey H5N1 Influenza Formulation C2 Group (N=40) | A/Turkey H5N1 Influenza Formulation D1 Group (N=61) | A/Turkey H5N1 Influenza Formulation D2 Group (N=46) | A/Turkey H5N1 Influenza Formulation E1 Group (N=59) | A/Turkey H5N1 Influenza Formulation E2 Group (N=41)
Pain (General disorders) | 41 | 59 | 9/40 | 53 | 10 | 48/60 | 13 | 46/58 | 6
Redness (General disorders) | 1 | 3 | 0/40 | 4 | 0 | 4/60 | 0 | 1/58 | 0
Swelling (General disorders) | 6 | 2 | 0/40 | 4 | 0 | 5/60 | 1 | 2/58 | 0
Fatigue (General disorders) | 10 | 18 | 3/40 | 20 | 6 | 18/60 | 4 | 23/58 | 11
Headache (General disorders) | 11 | 22 | 4/40 | 25 | 5 | 17/60 | 8 | 17/58 | 10
Joint pain (Infections and infestations) | 5 | 16 | 1/40 | 10 | 4 | 12/60 | 2 | 19/58 | 4
Muscle aches (General disorders) | 10 | 29 | 3/40 | 17 | 7 | 21/60 | 8 | 28/58 | 8
Shivering (General disorders) | 3 | 9 | 1/40 | 8 | 0 | 7/60 | 1 | 9/58 | 2
Sweating (General disorders) | 4 | 4 | 0/40 | 5 | 0 | 3/60 | 1 | 6/58 | 2
Fever (General disorders) | 0 | 1 | 0/40 | 0 | 0 | 4/60 | 0 | 4/58 | 0
Headache (Nervous system disorders) | 3 | 4 | 0 | 1 | 1 | 6 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 3 | 0 | 5 | 1 | 2 | 1 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 1 | 2 | 3 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 4
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.